CLINICAL TRIAL: NCT04894734
Title: The Feasibility of Epidural Electrical Stimulation (EES) for Improving Pain and Rehabilitation Outcomes in Patients With Spinal Cord Injury (SCI)
Brief Title: Spinal Cord Stimulation (SCS) for Spinal Cord Injury (SCI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nandan Lad, M.D., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Nandan Lad, M.D., Ph.D., Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00106738
Record Dates: First submitted 2021-05-07; First posted 2021-05-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injury at T1-T12 Level; Traumatic Thoracic Spinal Cord Contusion; Thoracic Spinal Cord Trauma; Traumatic Thoracic Spinal Cord Laceration; Post-Traumatic Thoracic Myelopathy; Traumatic Thoracic Spinal Cord Myelopathy
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EES on (Experimental): Patients will undergo epidural electrical stimulation (EES) and be allocated 1:1 to EES on.The patient and their family will be formally blinded to treatment assignment. The provider, research team, biostatistician and programming team will be unblinded to treatment assignments.
  Interventions: Device: EES on
- EES off (Placebo Comparator): Patients will undergo epidural electrical stimulation (EES) and allocated 1:1 to EES off.The patient and their family will be formally blinded to treatment assignment. The provider, research team, biostatistician and programming team will be unblinded to treatment assignments. Those in the EES off category will have their EES turned on at the 9-month time point.
  Interventions: Device: EES off

INTERVENTIONS:
Device: EES on — Epidural electrical stimulation (EES), also known as spinal cord stimulation (SCS), is a common FDA-approved therapy for chronic neuropathic pain of trunk and limb.
  Other Names: SCS (Spinal Cord Stimulation)
  Arms: EES on
Device: EES off — Epidural electrical stimulation (EES), also known as spinal cord stimulation (SCS), is a common FDA-approved therapy for chronic neuropathic pain of trunk and limb.
  Other Names: SCS
  Arms: EES off

SUMMARY:
The purpose of this feasibility study is to compare the impact of Spinal cord stimulation [SCS] for Spinal Cord Injury (SCI) pain and rehabilitation. SCS, also known as Epidural Electrical Stimulation (EES), will be utilized along with conventional medical management (CMM) or CMM alone. Participation in this research study is expected to last approximately 24 months. All subjects will be evaluated and proceed with implantation of two SCS devices- one tailored based on the individual's SCI for the treatment of neuropathic pain of trunk and limb and a second near the bottom of the spinal cord (conus region) to study the impact on motor, sensory, bowel/bladder outcomes. All patients will also continue receiving CMM, such as medications and physical therapy.

Participating subjects will be allocated to one of two treatment groups:

1. Placebo arm: SCS OFF + CMM. Under the direction of the study physician, the patient may receive a variety of treatments, such as medications and various forms of rehabilitation.
2. Treatment arm: SCS ON + CMM. The study treatment Spinal Cord Stimulation [SCS]: the study physician will perform a trial procedure to see if the study procedure works for the patient and may implant a permanent device if it is successful. There is a temporary trial procedure, or a "test drive," which usually lasts 5-7 days. If this is successful, patients will discuss a more permanent implant. This study involves the concurrent placement of two SCS devices (one focused on pain and the second for rehabilitation).

For three months, treatment group subjects will have the SCS turned on and will have rehabilitation as part of their CMM. Participants in the placebo arm will have their SCS remain off and will undergo CMM with rehabilitation therapy similar to the treatment group. Neither the subjects nor the treatment team will know which patients are in the treatment or placebo arm.

At the end of three months, the study group will be revealed and the placebo group subjects will be allowed to crossover and have their SCS turned on. Rehabilitation visits may be remote and the study duration is approximately 24 months. There may be additional blood tests and clinical exams to collect data on the effectiveness of the therapy. Data at follow-up visits will be compared to the subjects' baseline data and that of the control group at the respective visits.

DETAILED DESCRIPTION:
This study is a prospective, single center study. Data will be collected at baseline, time of procedure (trial and permanent), trial phase, and at 1, 3, 6, 12, 18, and 24 months post-implantation.

The primary objective of this study is to to determine if neuromodulation can be used to augment pain relief and rehabilitation in spinal cord injury (SCI) in a real-world population while further characterizing neurophysiological measures and clinical outcomes.

The following data will be collected:

* Medical history and demographics
* Procedure characteristics
* Medications
* Visual Analog Scale (VAS) for pain intensity Guy/Farrar Patient Global Impression of Change (PGIC) scale ASIA motor and sensory scores and impairment grade
* QoL survey (PROMIS 29)
* Electromyography (EMG) / Nerve Conduction Studies (NCS)
* Spinal Cord Independence Measure (SCIM) survey
* Bladder control using standard clinical urodynamic studies
* For sleep, self-reported quality and average hours per night will be collected in a diary
* Programming parameters and characteristics
* Safety events (adverse events, device deficiencies, protocol deviations)

The outcome variables of interest will be collected and assessed across study visits. No pre-planned formal statistical hypothesis tests will be performed. Multivariable regression modeling and descriptive statistics will be utilized.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study must meet all of the following inclusion criteria (based on investigator judgement):

1. Traumatic, thoracic SCI
2. Chronic neuropathic pain (i.e., Pain >3 for > 3 months)
3. Willing and able to provide informed consent, attend required study visits, and complete required assessments/questionnaires
4. 18-80 years of age
5. Medically stable enough to undergo surgical implantation of an SCS / participate in rehabilitation regimens

Exclusion Criteria:

Subjects enrolled in this study must not meet any of the following exclusion criteria (based on investigator judgement):

1. Complete cord transection
2. Persistent spinal instability or other injury preventing ability to participate
3. Active infection
4. Comorbid psychosis or psychotic disorder
5. Untreated, clinically significant depression
6. Active drug or alcohol abuse
7. Pregnant women or women who intend to become pregnant during the duration of the study. Women of childbearing potential need a negative pregnancy test
8. Patients without symptoms of neuropathic pain >3/10 for > 3 months
9. Patient deemed not medically stable for surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Multidimensional Pain Inventory (MPI)-SCI average activity score | Baseline, 3 months
  The MPI-SCI consists of twelve 7-point subscales in three sections: (1) pain impact, (2) responses by significant others, and (3) activity. Our primary outcome is the average score of the 4 pain subscales (household activities, activities away from home, social activities, and outdoor work) for pain and consequences of SCI. These 4 scales are commonly used to create a single general activity scale. To define the degree to which pain and other consequences of injury reduced participation in a specific activity, 2 additional validated items will be used in section 3: (1) "Pain has reduced my participation in this activity," and (2) "Other consequences of SCI have reduced my participation in this activity." The response range from 0 (not at all) to 6 (extremely).

SECONDARY OUTCOMES:
Change in pain as measured by Visual Analog Scales (VAS) | Baseline, and then months 1, 3, 6, 9, 12, 18 and 24
  Validated assessment of pain severity (0-10 scale), 0 being no pain to 10 being the worst pain, in the past 7 days.
Change in Quality of Life (QOL) as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 | Baseline, and then months 1, 3, 6, 9, 12, 18 and 24
  The PROMIS-29 is a generic health-related quality of life survey that assesses each of the 7 PROMIS domains with 4 questions. The questions are ranked on a 5-point Likert Scale. PROMIS instruments contain a fixed number of items from seven PROMIS domains: depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities. The seven domains cover the most relevant areas of self-reported health for the greatest majority of people with chronic illness.
Change in the overall improvement as measured by Guy/Farrar Patient Global Impression of Change (PGIC) scale | Baseline, and then months 1, 3, 6, 9, 12, 18 and 24
  The self-report measure PGIC reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement.
Change in motor recovery as measured by the Total American Spinal Injury Association (ASIA) motor score | Baseline, and then months 1, 3, 6, 9, 12, 18 and 24
  ASIA Upper Extremity and Lower Extremity Motor Score (UEMS & LEMS), combine to give Total ASIA Motor Score.
Change in motor recovery as measured by the ASIA impairment grades | Baseline, and then months 1, 3, 6, 9, 12, 18 and 24
  The ASIA Impairment Scale (AIS), based on the Frankel scale, is a clinician-administered scale used to classify the severity (completeness) of injury in individuals with SCI. It identifies sensory and motor levels indicative of the highest spinal level demonstrating "unimpaired" function. Preservation of function in the sacral segments (S4-S5) is a key for determining the AIS grade. AIS scores are considered essential when classifying persons with SCI as to their neurological status.
Change in independence of activities of daily living (ADLs) as measured by the Spinal Cord Independence Measure (SCIM) survey | Baseline, and then months 1, 3, 6, 9, 12, 18 and 24
  SCIM Disability scale developed to specifically address the ability of SCI patients to perform basic activities of daily living independently. Three versions of the SCIM (I-III) have been consecutively developed and assess three areas: 1) self-care (feeding, grooming, bathing, and dressing); 2) respiration and sphincter management; 3) mobility (bed and transfers and indoor/outdoor). The item scores are weighted related to the assumed clinical relevance.
Change in bladder control using urodynamics | Baseline, and then months 1, 3, 6, 9, 12, 18 and 24
  A urodynamic test is used to measure nerve and muscle function, pressure around and in the bladder, flow rates, and other factors. These tests look at how well the bladder, sphincters, and urethra are storing and releasing urine. All measures are combined to give one overall score of bladder control.
Change in motor recovery as measured by Transcranial Magnetic Stimulation Motor Evoked Potentials (TMS MEPs) | Baseline, and then months 1, 3, 6, 9, 12, 18 and 24
  To evaluate the connectivity of descending motor signals passing through the injury, TMS MEPs are recorded bilaterally over the rectus femoris (RF), vastus lateralis (VL), medial hamstring (MH), tibialis anterior (TA), medial gastrocnemius (MG), and soleus (SOL) muscles using skin surface EMG at a sampling rate of 4 kHz.
Change in motor recovery as measured by EMG | Baseline, and then months 1, 3, 6, 9, 12, 18 and 24
  EMGs will be recorded using surface or needle electrodes placed over/in the following muscles: bilateral gluteus maximus, bilateral rectus femoris, bilateral vastus lateralis, bilateral medial hamstrings, bilateral anterior tibialis and bilateral gastrocnemius. When clinically appropriate, bilateral extensor carpi radialis, bilateral biceps, and bilateral abdominal muscles will be used as controls.

CONTACTS AND LOCATIONS:
Overall Officials: Shivanand Lad, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473